CLINICAL TRIAL: NCT00919035
Title: Phase II Study Investigating the Toxicity and Efficacy of Single Agent Temsirolimus (Torisel®) in Chemotherapy-naïve Castration-Resistant Prostate Cancer Patients
Brief Title: Single Agent Temsirolimus (Torisel®) in Chemotherapy-naïve Castration-Resistant Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Director of Research, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSRI 0901
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; androgen-independent prostate cancer (AIPC) Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Torisel (Experimental): Single Agent Temsirolimus (Torisel®)
  Interventions: Drug: torisel

INTERVENTIONS:
Drug: torisel — Patients will receive Torisel 25 mg weekly. Treatment continues until disease progression, patient's withdrawal, unacceptable toxicity or the investigator's discretion
  Other Names: Temsirolimus

SUMMARY:
This is a single institution, open label, phase II study in androgen-independent prostate cancer patients who are chemotherapy-naïve. Patients will receive Torisel® 25 mg weekly. Treatment continues until disease progression, patient's withdrawal, unacceptable toxicity or the investigator's discretion.

DETAILED DESCRIPTION:
This is an open label phase II study conducted in patients who have androgen-independent and castration-resistant prostate cancer but who have not received systemic chemotherapy. Investigational therapy such as vaccines, immunotherapy, and some oral targeted agents are NOT considered chemotherapy. Prior use of steroids is not an exclusion criterion.

Patients who meet the inclusion criteria will be allowed to participate. Enrolled patients will receive single agent Torisel® at 25 mg weekly. Every 4 weeks of therapy will constitute one cycle of treatment. Patients will continue on therapy until voluntary withdrawal, toxicity, progression, or the investigator's discretion. Patients will be followed for 3 years after discontinuation of Torisel®.

Patients are allowed to receive intravenous or oral bisphosphonates for their bone metastases and are advised to continue androgen blockade while on study.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Documented prostate cancer regardless of the Gleason score
5. Patients should be considered hormone refractory and castration-resistant. They must fail LHRH analogues, and anti-androgen withdrawal trial. Failure is confirmed by an increase in PSA value of 10% or more than the value immediately before.
6. Patients must have measurable disease either biochemically (using PSA) and/or using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria for visceral organ involvement and/or bone disease. If there is no disease to follow on scans a PSA value of at least 5 ng per milliliter needs to be present at baseline to be evaluated for PSA response.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or less.
8. Adequate liver function tests with ALT/AST being < 3x normal, total bilirubin of 1.5 or less, and adequate renal function measured by a creatinine of 2.0 mg/dl or less. Alkaline phosphatase values are never exclusion criteria if it is deemed related to bone metastases.
9. Patients need to have adequate bone marrow function.

   * absolute neutrophil count (ANC) of 1000 or above,
   * Hgb of 9.0 g/dl or above,
   * Platelets of 100,000 or above. If other causes are affecting plts counts such as autoimmune disorders, patients are allowed on study. Patients with inadequate bone marrow function that is deemed related to bone marrow involvement with prostate cancer (cytopenias are due to extensive marrow infiltration with prostate cancer) are allowed at the investigator's discretion.
10. Patients with other malignancies are allowed as long as there is no evidence of the other malignancy present at entry time, and it has been 3 years or more since the treatment for the other disorder was completed. Patients with non-melanoma skin cancers are allowed to participate in the study.
11. Investigational therapy such as vaccines, immunotherapy, and oral targeted agents are allowed on this study as long as their last exposure was 4 weeks prior to study entry. These agents are not considered an exclusion criteria as they are not considered standard chemotherapy.
12. Patients with known bone metastases are allowed to receive intravenous bisphosphonates such as aredia or zometa. Patients on oral bisphosphonates are also allowed.
13. All study participants are encouraged to continue androgen deprivation with an LHRH analogue.
14. Patients must agree to use a latex condom during sexual contact with a female of childbearing potential, even if they have had a successful vasectomy and despite the fact that they are on androgen deprivation.
15. Last treatment for prostate cancer should be at least 4 weeks ago

Exclusion Criteria:

1. Prior systemic chemotherapy for castration Resistant Prostate Cancer (CRPC)
2. Prior exposure to temsirolimus (TEM)
3. Known HIV positive status or infectious hepatitis, type A, B, or C.
4. Known brain metastases.
5. Steroids are allowed concomitantly ONLY IF they are taken for another chronic medical condition (Such as chronic obstructive pulmonary disease , Multiple sclerosis…etc)
6. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing and understanding the informed consent form.
7. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study or confounds the ability to interpret data from the study.
8. Use of any other experimental drug or therapy within 28 days of baseline.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-06; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, S.C.
Locations (2):
- United States (2):
  - Oncology Specialists, SC, Niles, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Torisel
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Torisel: Single Agent Temsorilmus (Torisel®)
  Patients will receive Torisel 25 mg weekly given as an intravenous infusion on days 1, 8, 15 and 33 every 28 days. Treatment continues until disease progression, patient's withdrawal, unacceptable toxicity or the investigator's discretion
Arm/Group | Torisel
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Benefit From Torisel® in Chemotherapy-naïve Castration Resistant Prostate Cancer (CRPC).
Description: The overall clinical benefit is defined as the sum of complete response (CR), partial response (PR), and stable disease (SD). CR: is the disappearance of all measurable lesions including bone lesions detected on the bone scan, no evidence of new lesions, and no disease-related symptoms. PR: More than 30% decrease in the sum of longest diameter of measurable lesions compared to baseline. SD: Lesions should have no sufficient decrease for PR or CR and no sufficient increase to meet criteria for Progressive Disease (PD). PD: > 20% increase in the sum of longest diameter of measurable lesions compared to baseline, and/or evidence of new lesions on imaging studies OR The appearance of 2 or more new bony lesions on a bone scan is satisfactory for PD. Newly developed cord compression or pathologic fracture is defined as PD.
Time Frame: disease progression is assessed every 2 cycles, for up to 40weeks, per protocol, from the date of the first dose of study drug to the date the patient is taken off study
Measure: Number; unit: percentage of participants
Groups:
- Torisel: Single Agent Temsirolimus (Torisel®)
  Patients will receive Torisel 25 mg weekly given as an intravenous infusion on days 1, 8, 15 and 33 every 28 days. Treatment continues until disease progression, patient's withdrawal, unacceptable toxicity or the investigator's discretion
Arm/Group | Torisel
Number analyzed (Participants) | 15
percentage of participants | 67

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the length of time from when the patient starts the study till disease progression. Disease progression is defined as more than 20% increase in the sum of longest diameter of measurable lesions compared to baseline, and/or evidence of new lesions on imaging studies. Or the appearance of 2 or more new bony lesions on a bone scan. Or newly developed cord compression or pathologic fracture.
Time Frame: Disease progression is assessed every 2 months, for up to 40 weeks, measured from day one of protocol treatment until the date the patient is off study.
Measure: Mean (Full Range); unit: months
Arm/Group | Torisel
Number analyzed (Participants) | 15
months | 2 [2 to 10]

3. Secondary Outcome: Does the Prostate Specific Antigen (PSA) Doubling Times Change Before and After Treatment
Description: PSA Doubling time is defined as the length of time that it takes for an individual patients PSA to double. PSA doubling times were calculated using the medial records at study entry for each patient. While the patient was on study their PSA doubling times were also calculated.
Time Frame: evaluate PSA doubling time pre study to actual doubling time while on study - calculated from start of study up to 10 cycles or 40 weeks.
Population: PSA doubling time pre study was compared to PSA doubling time while the patients are on study, per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Torisel
Number analyzed (Participants) | 14
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the start of the study until study completion. This is from May 2009 until October 2013.
Arm/Group | Torisel
Serious Adverse Events (participants affected / at risk) | 11/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Torisel (N=21)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Acute Arterial ischemia (Vascular disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
fever (Infections and infestations) | 1 (1)
intracranial bleed (Vascular disorders) | 1 (1)
pain (General disorders) | 4 (4)
pneumonia (General disorders) | 3 (3)
renal failure (Renal and urinary disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
transient ischemic attack (Vascular disorders) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 2 (2)
weakness (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Torisel (N=21)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
anxiety (Psychiatric disorders) | 5 (5)
albumin low (Metabolism and nutrition disorders) | 8 (8)
anemia (Blood and lymphatic system disorders) | 15 (15)
anorexia (Metabolism and nutrition disorders) | 11 (11)
alkaline phosphatase (General disorders) | 6 (6)
Aspartate Aminotransferase elevated (General disorders) | 8 (8)
Alanine Aminotransferase high (General disorders) | 2 (2)
bruising (Vascular disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
creatinine high (Renal and urinary disorders) | 7 (7)
constipation (Gastrointestinal disorders) | 9 (9)
chills (General disorders) | 2 (2)
depression (Psychiatric disorders) | 6 (6)
dehydration (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
eyes dry (Eye disorders) | 2 (2)
eyes watery (Eye disorders) | 3 (3)
edema (Vascular disorders) | 7 (7)
fall (General disorders) | 2 (2)
fatigue (General disorders) | 15 (15)
fever (Infections and infestations) | 2 (2)
gynecomastia (General disorders) | 2 (2)
hypercholesteremia (General disorders) | 8 (8)
hypercalcemia (General disorders) | 3 (3)
hyperglycemia (General disorders) | 14 (14)
hypertriglyceridemia (General disorders) | 14 (14)
hematuria (Renal and urinary disorders) | 2 (2)
hypoglycemia (General disorders) | 1 (1)
hypocalcemia (General disorders) | 9 (9)
hypokalemia (General disorders) | 5 (5)
hyponatremia (General disorders) | 6 (6)
hypophosphatemia (General disorders) | 5 (5)
hemorrhoids (General disorders) | 2 (2)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
infection (Infections and infestations) | 2 (2)
insomnia (General disorders) | 3 (3)
lightheadedness (General disorders) | 1 (1)
leukopenia (General disorders) | 15 (15)
lymphopenia (General disorders) | 13 (13)
mucositis (General disorders) | 5 (5)
neutropenia (General disorders) | 12 (12)
neuropathy (Nervous system disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 4 (4)
protein low (Metabolism and nutrition disorders) | 2 (2)
pain (General disorders) | 8 (8)
rash (Skin and subcutaneous tissue disorders) | 7 (7)
rectal fissure (General disorders) | 2 (2)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
taste changes (Metabolism and nutrition disorders) | 3 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)
vomting (Gastrointestinal disorders) | 3 (3)
weight loss (General disorders) | 6 (6)
weakness (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No